CLINICAL TRIAL: NCT01052025
Title: Antiatherogenic and Antimetabolic Effect of Curcumin Therapy in the Prevention and Delay of Type 2 Diabetic in Patients With Impaired Glucose Tolerance and Insulin Resistance
Brief Title: Curcumin Therapy in Patients With Impaired Glucose Tolerance and Insulin Resistance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Srinakharinwirot University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Assit.Prof. Somlak Chuengsamarn, Department of Internal Medicines, Faculty of Medicine, Srinakarinwirot University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SWUEC9/2552
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-03

CONDITIONS: Type 2 Diabetes; Pre-diabetes; Insulin Resistance; Cardiovascular Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Insulin Resistance | interventions — Curcumin; Tacrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin (Experimental): curcumin capsule contains 250 mg curcuminoiods, 3 capsules per time, 2 times a day before meal for 12 months
  Interventions: Drug: Curcumin
- Placebo (No Intervention)

INTERVENTIONS:
Drug: Curcumin — curcumin capsule contains 250 mg curcuminoiods, 3 capsules per time, 2 times a day before meal for 12 months
  Other Names: Curcumin capsules are manufactured by Government Pharmaceutical Organization, Thailand
  Arms: Curcumin

SUMMARY:
The incidence rate of type 2 diabetes in Thai populations is high and increasing every year. Cardiovascular disease is the main complication of this disease, which has been defined as an important cause of death among Diabetic patients. This disease is now becoming a major health problem and causes a great economic loss to the country. Evidence shows that Curcumin, Thai herbal medicine, has the effectiveness of prevention and delay of type 2 diabetes. However, there is no scientific study that aims to prove the efficacy of this herb particularly for prevention and delay the disease in Patients with impaired glucose tolerance (pre-diabetes) and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35 years or older with an abnormal fasting plasma glucose (100-125 mg/dl) or with insulin resistance (140-199 mg/dl) by using 75 mg of glucose OGTT.

Exclusion Criteria:

* Have been diagnosed with diabetes by the results of FPG >/=126 mg/dl
* Present with secondary peripheral arterial disease (PAD)
* Present with cardiovascular diseases such as coronary arterial disease and cerebrovascular disease
* Receive anticoagulant drugs that have an effect on the measurement of pulse wave velocity (PWV)
* Receive antihypertensive or lipid-lowering drugs (ARB, ACEI, fenofibrate, atorvastatin, rosuvastatin, fluvastatin) that have an effect on the measurement of C-reactive protein (CRP)
* Present with kidney failure (serum creatinine > 2.0 mg/dl) or in the process of renal dialysis
* Present with hepatitis (ALT level >/= 3 times the upper limit)
* Receive any herbal medications or curcumin
* Present with high blood sugar from other causes apart from type 2 diabetes such as receiving steroid drugs, cancer or pancreatic cyst
* Present with infection or inflammation that have effect on the level of CRP
* Pregnancy or breastfeeding
* Have a history of gall bladder diseases or removal

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To examine the efficacy of curcumin on the delay of degenerative beta-cells in pancrease for protection of Type 2 Diabetes in patients with impaired glucose tolerance (Pre-diabetes) | 12 months

SECONDARY OUTCOMES:
To examine the efficacy of curcumin on the reduction of blood sugar level, lipid profile, insulin resistance status and oxidative stress status in Pre-diabetes patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Somlak Chuengsamarn, Medical Doctor, Principal Investigator — Srinakarinwirot University
Locations (1):
- HRH Princess Maha Chakri Sirindhorn Medical Center, Ongkarak, Nakornnayok, Thailand

REFERENCES:
- [Derived] Chuengsamarn S, Rattanamongkolgul S, Luechapudiporn R, Phisalaphong C, Jirawatnotai S. Curcumin extract for prevention of type 2 diabetes. Diabetes Care. 2012 Nov;35(11):2121-7. doi: 10.2337/dc12-0116. Epub 2012 Jul 6. PMID 22773702